CLINICAL TRIAL: NCT01185847
Title: A Randomized, Multicenter, Open-label Phase Ib/II Study of RO5083945 in Combination With Cisplatin and Gemcitabine/Pemetrexed Versus Cisplatin and Gemcitabine/Pemetrexed in Patients With Advanced or Recurrent Non Small Cell Lung Cancer Who Have Not Received Prior Chemotherapy
Brief Title: A Study of RO5083945 in Combination With Chemotherapy Versus Chemotherapy Alone in Patients With Advanced or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP22349; 2010-018945-72
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — imgatuzumab; Cisplatin; Gemcitabine; Pemetrexed

ARMS (4):
- A non-squamous (Experimental)
  Interventions: Drug: RO5083945; Drug: cisplatin; Drug: pemetrexed
- A squamous (Experimental)
  Interventions: Drug: RO5083945; Drug: cisplatin; Drug: gemcitabine
- B non-squamous (Active Comparator)
  Interventions: Drug: cisplatin; Drug: pemetrexed
- B squamous (Active Comparator)
  Interventions: Drug: cisplatin; Drug: gemcitabine

INTERVENTIONS:
Drug: RO5083945 — intravenously, until disease progression
  Arms: A non-squamous; A squamous
Drug: cisplatin — standard treatment, up to 6 cycles
Drug: gemcitabine — standard treatment, up to 6 cycles
  Arms: A squamous; B squamous
Drug: pemetrexed — standard treatment, up to 6 cycles
  Arms: A non-squamous; B non-squamous

SUMMARY:
This open label, 2-part study will evaluate the safety and efficacy of RO5083945 in combination with standard chemotherapy in patients with advanced or recurrent non-small cell lung cancer who have not received prior chemotherapy. In Part 1 patients will receive RO5083945 intravenously and standard chemotherapy (cisplatin plus either gemcitabine or pemetrexed) for up to 6 cycles of 3 weeks and then RO5083945 until disease progression. In Part 2 patients will be randomized to receive either RO5083945 in combination with standard chemotherapy or chemotherapy alone for up to 6 cycles. In the absence of disease progression, patients receiving RO503945 can continue treatment with RO5083945 as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Advanced (IIIb), metastatic (IV) or recurrent non-small cell lung cancer
* At least 1 measurable disease lesion as per RECIST criteria
* Confirmed presence of EGFR in tumor tissue
* ECOG performance status 0-1
* Adequate hematological, renal and liver function

Exclusion Criteria:

* Prior chemotherapy or treatment with another systemic anti-cancer agent
* Radiotherapy within the last 4 weeks, except for limited field palliative radiotherapy for bone pain relief
* Symptomatic or active CNS metastases
* Recent history of poorly controlled hypertension (systolic >180mmHg or diastolic >100mmHg)
* Requirement for steroids > 40 mg prednisolone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Part 2: Progression-free survival, according to RECIST criteria by CT/MRI | 23 months
Part 1: Adverse event profile: adverse events, ECG, hematology, urinalysis, human anti-human antibodies (HAHA) | 6 months

SECONDARY OUTCOMES:
Pharmacokinetics of RO5083945 (AUC, Cmax and Cmin) in combination with cisplatin and gemcitabine/pemetrexed | multiple sampling cycles 1-6 (18 weeks)
Duration of response, according to RECIST criteria by CT/MRI | from response to disease progression
Clinical benefit rate (complete response, partial response or stable disease for >/=6 weeks), according to RECIST criteria by CT/MRI | 23 months
Overall survival | 23 months
Overall response rate (ORR), according to RECIST criteria by CT/MRI | 23 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- Belgium (3):
  - Charleroi
  - Leuven
  - Liège
- France (4):
  - Caen
  - Marseille
  - Saint-Herblain
  - Toulouse
- Germany (7):
  - Bad Berka
  - Cologne
  - Gauting
  - Großhansdorf
  - Heidelberg
  - Mainz
  - Mannheim
- Italy (5):
  - Milan, Lombardy
  - Ancona, The Marches
  - Lido di Camaiore, Tuscany
  - Livorno, Tuscany
  - Perugia, Umbria
- Poland (3):
  - Lodz
  - Otwock
  - Warsaw
- Spain (4):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Málaga, Malaga
  - Seville, Sevilla
- London, United Kingdom